CLINICAL TRIAL: NCT00932204
Title: A Randomized, Controlled Study of Sequentially Applied Repetitive Transcranial Magnetic Stimulation in Obsessive- Compulsive Disorders
Brief Title: Study of Sequentially Applied Repetitive Transcranial Magnetic Stimulation in Obsessive- Compulsive Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Se Joo Kim, Professor, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2006-0318
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Obsessive-compulsive Disorder
Keywords: obsessive-compulsive disorder; repetitive transcranial magnetic stimulation; right dorsolateral prefrontal cortex; supplementary motor area (SMA)
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active stimulation (Experimental): For the active group, rTMS over the right prefrontal cortex and the SMA was sequentially performed. The rTMS of the right dorsolateral prefrontal cortex was conducted at a point 5 cm anterior to the point at which the MT was determined, and it was administered at an intensity of 110% of the RMT, a frequency of 1 Hz, for 10 minutes, and with an inter-train interval of 2 minutes (1200 stimuli/d).
  The vertex (Cz) was measured for each patient, and the SMA was defined at 15% of the distance between the inion and nasion anterior to Cz on the sagittal midline, according to the international 10-20 EEG system. The rTMS over the SMA was administered at an intensity of 100% of the RMT, a frequency of 1 Hz, for 10 minutes and with an inter-train interval of 2 minutes (1200 stimuli/d).
  Interventions: Device: repetitive transcranial magnetic stimulation (Magstim rapid magnetic stimulator)
- Sham stimulation (Sham Comparator): For the sham group, the sham stimulation was applied with the coil angled at 45° from the scalp using the same parameters as the active stimulation group over the same area.
  Interventions: Device: repetitive transcranial magnetic stimulation (Magstim rapid magnetic stimulator)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (Magstim rapid magnetic stimulator) — For the active group, rTMS over the right prefrontal cortex and the SMA was sequentially performed. The rTMS of the right dorsolateral prefrontal cortex was conducted at a point 5 cm anterior to the point at which the MT was determined, and it was administered at an intensity of 110% of the RMT, a frequency of 1 Hz, for 10 minutes, and with an inter-train interval of 2 minutes (1200 stimuli/d).
  The vertex (Cz) was measured for each patient, and the SMA was defined at 15% of the distance between the inion and nasion anterior to Cz on the sagittal midline, according to the international 10-20 EEG system. The rTMS over the SMA was administered at an intensity of 100% of the RMT, a frequency of 1 Hz, for 10 minutes and with an inter-train interval of 2 minutes (1200 stimuli/d).
  For the sham group, the sham stimulation was applied with the coil angled at 45° from the scalp using the same parameters as the active stimulation group over the same area.
  Other Names: A Magstim rapid magnetic stimulator with a 70-mm figure-of-eight coil (Magstim Company Ltd, Whitland, UK) was used for treatment.

SUMMARY:
The purpose of study was to investigate possible therapeutic effects and safety of sequentially combined low-frequency repetitive transcranial magnetic stimulation (rTMS) to the right dorsolateral prefrontal cortex (DLPFC) and supplementary motor area (SMA) in patients with treatment-resistant obsessive-compulsive disorder (OCD).

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a relatively common psychiatric disorder characterized by repetitive, intrusive thoughts and time-consuming behavioral or mental acts. Many OCD patients who do not respond to conventional treatments experience severe distress and disruptions in their daily activities. Novel approaches including psychopharmacological therapy and surgical techniques for treatment-resistant OCD have been proposed. With recent advances in non-invasive technique for stimulating the cerebral cortex, repetitive transcranial magnetic stimulation (rTMS) has been proposed as a potential therapeutic approach for various psychiatric illnesses including OCD.

Because of contradictory findings and a lack of controlled trials in OCD, rTMS cannot be yet recommended as routine therapy for OCD. However, it may have a potential clinical effect as a putative add-on treatment for OCD and an alternative therapy for treatment-resistant OCD.

For useful clinical applications, it is very important to develop methods to enhance the efficacy of rTMS. There are a number of putative ways to do this, and one of them is sequentially combining two forms of stimulation which are considered to have potential therapeutic effects. More recently, the sequential application of two stimulation regimens (high-frequency left-side rTMS and low-frequency right-side rTMS to the prefrontal cortex) has been found to have a substantial therapeutic effect in patients with treatment-resistant major depression. Therefore, the investigation for a sequentially combining effect of both the right prefrontal and the SMA stimulation would be worthwhile in OCD patients.

ELIGIBILITY:
Inclusion Criteria:

* OCD patients who had failed adequate trials (a lack of at least a 25% reduction in the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) 15 after at least eight weeks of treatment) of at least two serotonin re-uptake inhibitors (SRI) and behavioral therapy.

Exclusion Criteria:

* Subjects were excluded if:

  * they presented with a movement disorder other than a tic
  * any psychotic symptoms
  * other anxiety disorders
  * mental retardation
  * alcohol or other substance abuse within the last six months
  * a history of psychosurgery, encephalitis or significant head trauma

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2007-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for the study was score on the Y-BOCS. The responder on Y-BOCS is defined as a Y-BOCS decrease at least 25% from the baseline at post-treatment (at 4 weeks) | baseline, week 1, week 2, and week 4

SECONDARY OUTCOMES:
The secondary outcome measures were the scores of MADRS and HARS, to examine the effects on cognitive functions of rTMS, a computerized Stroop task was conducted and side effect checklist. | baseline, week 1, week 2, and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Se Joo Kim, M.D., Principal Investigator — Yonsei Univ. College of Medicine
Locations (1):
- Yonsei Univ. Health System Severance Hospital, Seoul, South Korea

REFERENCES:
- [Result] Mantovani A, Lisanby SH, Pieraccini F, Ulivelli M, Castrogiovanni P, Rossi S. Repetitive transcranial magnetic stimulation (rTMS) in the treatment of obsessive-compulsive disorder (OCD) and Tourette's syndrome (TS). Int J Neuropsychopharmacol. 2006 Feb;9(1):95-100. doi: 10.1017/S1461145705005729. Epub 2005 Jun 28. PMID 15982444
- [Result] Sachdev PS, McBride R, Loo CK, Mitchell PB, Malhi GS, Croker VM. Right versus left prefrontal transcranial magnetic stimulation for obsessive-compulsive disorder: a preliminary investigation. J Clin Psychiatry. 2001 Dec;62(12):981-4. doi: 10.4088/jcp.v62n1211. PMID 11780880
- [Derived] Kang JI, Kim CH, Namkoong K, Lee CI, Kim SJ. A randomized controlled study of sequentially applied repetitive transcranial magnetic stimulation in obsessive-compulsive disorder. J Clin Psychiatry. 2009 Dec;70(12):1645-51. doi: 10.4088/JCP.08m04500. Epub 2009 Aug 25. PMID 19709504